CLINICAL TRIAL: NCT06647251
Title: Comparison of 3 RF Delivery Modes of the QDOT Catheter for Paroxymal AF Ablation: a Prospective Study
Brief Title: Comparison of 3 RF Delivery Modes of the QDOT Catheter for Paroxymal Atrial Fibrillation (AF) Ablation
Acronym: QDOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RYTHMO-03-2024
Record Dates: First submitted 2024-08-27; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of the following arms: Q-MODE, Q-MODE+, hybride Q-MODE/Q-MODE+.
  The number of patients in each arm is the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Q-MODE (Active Comparator): Radiofrequency ablation with High Power - Short Duration (HPSD) up to 50W.
  Interventions: Procedure: Q-MODE : radiofrequency ablation up to 50W
- Q-MODE+ (Active Comparator): Radiofrequency ablation with High Power - Short Duration (HPSD) up to 90W.
  Interventions: Procedure: Q-MODE+ : radiofrequency up to 90W
- Hybride Q-MODE/Q-MODE+ (Active Comparator): A combination of the two ablation methods.
  Interventions: Procedure: Hybride Q-MODE/Q-MODE+: radiofrequency ablation up to 50W in the anterior part, and 90W in the posterior part

INTERVENTIONS:
Procedure: Q-MODE : radiofrequency ablation up to 50W — The same device (QDOT Micro™) is used in all 3 arms of this trial. The 3 strategies of radiofrequency delivery within the 3 arms are already used in the standard of care.
  For patient randomized in this arm, the device is set to Q-MODE option: the intensity of radiofrequency to isolate the pulmonary vein is limited to 50W.
  Arms: Q-MODE
Procedure: Q-MODE+ : radiofrequency up to 90W — The same device (QDOT Micro™) is used in all 3 arms of this trial. The 3 strategies of radiofrequency delivery within the 3 arms are already used in the standard of care.
  For patient randomized in this arm, the device is set to Q-MODE+ option: the intensity of radiofrequency to isolate the pulmonary vein is limited to 90W.
  Arms: Q-MODE+
Procedure: Hybride Q-MODE/Q-MODE+: radiofrequency ablation up to 50W in the anterior part, and 90W in the posterior part — The same device (QDOT Micro™) is used in all 3 arms of this trial. The 3 strategies of radiofrequency delivery within the 3 arms are already used in the standard of care.
  For patient randomized in this arm, the device is set to "Q-MODE/Q-MODE+" option: the intensity of radiofrequency delivered to isolate the pulmonary vein is limited to 50W in the anterior part and to 90W in the posterior part.
  Arms: Hybride Q-MODE/Q-MODE+

SUMMARY:
Pulmonary vein isolation is the main treatment of paroxysmal and persistent atrial fibrillation.

The aim of our study is to prospectively compare the efficacy and safety of the 3 options of radiofrequency delivery with QDOT Micro™, with systematic use of catheter stabilization tools and tighter lesions

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) is the main treatment of paroxysmal and persistant atrial fibrillation.

PVI is achieved by point-by-point radiofrequency ablation that creates flexible lesion set within targeted area.

PVI using standard ablation catheter with limited power (50W) have been described in case series with favorable efficacy and safety.

QDOTMicro™ is a radiofrequency ablation catheter that incorporates advanced, high-energy ablation, improved temperature monitoring, optimized irrigation, and higher signal resolution.

QDOT Micro™ provides several options regarding radiofrequency administration :

* Q-MODE : provides high power short duration (HPSD) unitl 50W radiofrequency,
* Q-MODE+ : provides very high power very short duration (vHSPD) until 90W radiofrequency,
* Hybrid Q-MODE/Q-MODE+ : is a combination of two methods. In our experience, stability is a prerequisite for PVI with QDOT Micro™.

Small series have described encouraging results (85% isolation, unpublished data) with stabilization tools such as low-volume ventilation or apnea, high-rate simualtion, Vizigo bi-directional sheath (Vizigo™).

Recently, preliminary animal data argue in favor or reducing the interpoint distance with QDOT™.

To date, there is no study comparing the 3 options of radiofrequency delivery. The aim of our study is to prospectively compare the efficacity and safety of the 3 options of radiofrequency delivery with QDOT Micro™, with systematic use of catheter stabilization tools and tighter lesions.

The same device is used in all three randomisation groups. The difference between the intervention is the intensity of the radiofrequency applied.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* First atrial fibrillation ablation
* Paroxysmal atrial fibillation defined as atrial fibrillation lasting less than 48 hours
* Early atrial fibrillation defined as atrial fibrillation lastiing between 7 days and 3 months
* At least one episode of atrial fibrillation in the year preceding study entry
* Patient affiliated to a health insurance

Exclusion Criteria:

* History of atrial fibrillation ablation (surgery or catheter)
* Documented left atrial thrombus
* Left atrial (LA) diameter > 60mm / LA area > 35cm2 / Left atrial volulme index (LAVI) > 45ml/m2
* N/STEMI replacement or angioplasty or valve within 3 months prior to registration
* Any contraindication mentioned in the instructions for use of the QDOT MICRO™ bidirectional navigation catheter
* Patient unable to understand study information
* Patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of primary adverse events related to the ablation procedure | 7 days after ablation
  Incidence of primary adverse events within 7 days after ablation in the 3 arms
Acute procedural success | At the end of the ablation procedure
  Acute procedural success is defined as electrical isolation of all pulmonary veins

SECONDARY OUTCOMES:
Incidence of serious adverse event | within 7 days (early onset), 7 to 30 days (periprocedural), up to 18 months (late onset) of the ablation procedure
  Incidence of serious adverse events
Rate of additional lesions | At the end of the ablation procedure
  Rate of additional lesions between all targeted veins and per subject
Location of additional lesions | At the end of the ablation procedure
  Anatomical location of additional lesions
Use of another catheter | At the end of the ablation procedure
  Use of another catheter than QDOT in all targeted veins
Time spent in operating room | At the end of the ablation procedure
  Time spent in operating room
Skin-to-skin time | At the end of the ablation procedure
  Skin-to-skin time
Glove-to-glove time | At the end of the ablation procedure
  Glove-to-glove time = total procedure time
Mapping time | At the end of the ablation procedure
  Mapping time
Total ablation time | At the end of the ablation procedure
  Total ablation time
Left vein ablation time | At the end of the ablation procedure
  Left vein ablation time
Right vein ablation time | At the end of the ablation procedure
  Right vein ablation time
Number of radiofrequency applications | At the end of the ablation procedure
  Number of radiofrequency applications
Number of vHPSD radiofrequency applications | At the end of the ablation procedure
  Number of vHPSD (very High Power Short Duration) radiofrequency applications
Number of HPSD radiofrequency applications | At the end of the ablation procedure
  Number of HPSD (High Power Short Duration) radiofrequency applications
Temperature | At the end of the ablation procedure
  Temperature
Power | At the end of the ablation procedure
  Power
Contact force | At the end of the ablation procedure
  Contact force
Impedance | At the end of the ablation procedure
  Impedance

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric SEBAG, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, Paris, France